CLINICAL TRIAL: NCT02880384
Title: Projected Influence of Enhanced Pathogen Detection on the Clinical Management of Community-Acquired Pneumonia
Brief Title: Pathogen Detection and Community Acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-172A
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FilmArray LRTI v.2.0 IUO Panel (Experimental): Patients will provide sputum or sputum equivalent for FilmArray LRTI v.2.0 IUO Panel testing.
  Interventions: Other: FilmArray LRTI v.2.0 IUO Panel

INTERVENTIONS:
Other: FilmArray LRTI v.2.0 IUO Panel — Patients will provide sputum or sputum equivalent to be probed with FilmArray LRTI v.2.0 IUO Panelpanel.

SUMMARY:
Study to compare the number of community-acquired pneumonia (CAP) pathogens detected using current diagnostic tests to the number detected using the BioFire Diagnostics investigational polymerase chain reaction (PCR) platform.

DETAILED DESCRIPTION:
Patients diagnosed in the emergency department with CAP that requires hospitalization provide a sputum sample for culture and sensitivity testing, urine for detection of S. pneumonia and L. pneumophila, an anterior nasal swab for S. aureus PCR, a nasopharyngeal swab for S. pneumonia PCR and the FilmArray LRTI v.2.0 IUO Panel, and blood for procalcitonin testing and, in cases in which the patient is suffering rigors and hypotension, cultures. As part of this study, sputum or sputum equivalent will be acquired for testing using the FilmArray LRTI v.2.0 IUO Panel.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department physician diagnosis of CAP requiring hospitalization

Exclusion Criteria:

* Inability to obtain sputum or sputum equivalent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Pathogen Detection | 5 Days
  Compare the number of CAP pathogens detected using current diagnostic bundle to the number detected using the FilmArray LRTI v.2.0 IUO Panel.

SECONDARY OUTCOMES:
Treatment Influence | 5 Days
  Determine the number of cases in which the FilmArray LRTI v.2.0 IUO Panel could allow for a switch from empiric to specific antimicrobial therapy if the results had been known by the healthcare provider.
Nasopharyngeal swabs compared to sputum | 5 Days
  Compare the number of pathogens detected using an approved PCR panel using nasopharyngeal swabs to the number detected using the FilmArray LRTI v.2.0 IUO Panel.

CONTACTS AND LOCATIONS:
Overall Officials: David Gilbert, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Portland Providence Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No